CLINICAL TRIAL: NCT02328144
Title: Effectiveness of Metronidazole Versus Homologated Placebo in Pain Control Posthemorrhoidectomy
Brief Title: Effectiveness of Metronidazole in Pain Control Posthemorrhoidectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, CLOTILDE FUENTES OROZCO, PhD, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2013-1301-71
Record Dates: First submitted 2014-12-22; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoidectomy; Postoperative pain; Metronidazole
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metronidazole (Active Comparator): 22 patients received oral metronidazole 500mg 3 times for day for 7 days
  Interventions: Drug: Metronidazole
- Placebo (Placebo Comparator): 22 patients received oral placebo 500mg 3 times for day for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metronidazole — Patients were assigned to two groups, one of them received oral metronidazole (study group) and the other, homologated placebo (control group) after hemorrhoidectomy. Then, postoperative pain was assessed by visual analog scale at 6 and 12hrs, 1, 4, 7 and 14 days
  Other Names: Flagyl
  Arms: Metronidazole
Drug: Placebo — Patients were assigned to two groups, one of them received oral metronidazole (study group) and the other, homologated placebo (control group) after hemorrhoidectomy. Then, postoperative pain was assessed by visual analog scale at 6 and 12hrs, 1, 4, 7 and 14 days.
  Other Names: Homologated Placebo
  Arms: Placebo

SUMMARY:
Hemorrhoidal disease occurs in 50% of people over 40 years old and is the most common cause of anorectal surgery. One of the complications of hemorrhoidectomy is pain, which is a difficult symptom to appreciate and assess, by its frequent and large variations in sensitivity in each patient. Many studies have been done to reduce patient postoperative pain, but there is no ideal method. The application of both oral and topical metronidazole has shown to decrease pain following hemorrhoidectomy, but its use is not standardized.

The investigators evaluated the effect of oral administration of metronidazole versus homologated placebo in pain control after hemorrhoidectomy

DETAILED DESCRIPTION:
Objective: Evaluate the effect of oral administration of metronidazole versus homologated placebo in pain control after hemorrhoidectomy.

Material and methods: Controlled clinical trial, composed of 44 patients in a randomized manner, realized at the Coloproctology, Western Medical Center, Mexican Institute of Social Security. Referred beneficiaries adults were included, of either sex, who merited elective hemorrhoidectomy for hemorrhoidal disease grades III-IV using Ferguson's technique. They were assigned to receive metronidazole (study group) or homologated (control group) and the randomization was conducted by sealed envelopes and subsequently. We collected demographic and clinical variables. Postoperative pain was assessed by visual analog scale at 6 and 12hrs, 1, 4, 7 and 14 days; additional analgesic use; complications; return to normal activity and patient satisfaction; also were measured, in a blood sample after surgery and 12 hrs later, interleukin 6 and 10.

The statistical analysis was performed according to the nature of variables, for continuous data using measures of central tendency and dispersion and for the qualitative data with frequencies and percentages

ELIGIBILITY:
Inclusion Criteria:

* Hemorrhoidal disease grade III and IV
* Informed consent

Exclusion Criteria:

* Pregnancy
* Lactation
* Other anorectal disease
* Previous anorectal
* hypersensibility to metronidazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pain evolution, hours and days after surgery | 6 and 12 hours, 1, 4, 7 and 14 days
  Pain was assessed with the visual analogue scale questionnaire

SECONDARY OUTCOMES:
Interleukin | after surgery and 12 hours
  In a blood sample, right after surgery and 12 hours later, interleukin 6 and 10 were measured by ELISA, observing if they presented alterations with the intervention, between 2 groups and between the hours the investigators took the blood sample
Analgesics | 6 and 12 hours, 1, 4, 7 and 14 days
  Using a questionnaire if they used analgesics, which one, dose of it and how many days
Surgery complications | 6 and 12 hours, 1, 4, 7 and 14 days
  Asking directly to participants if they presented bleeding, urinary retention or another complication. Investigators measured how many participants presented complications
Return to normal activities | 1, 4, 7 and 14 days
  Asking to participans when they return to normal activities (to walk normally, to cook, to bath, to wear, to work) How many days were needed to recover their normal activities
Satisfaction | 14 day
  Asking how they felt in last 14 days and what was their perception of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde Fuentes-Orozco, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Western Medical Center, Mexican Institute of Social Security, Guadalajara, Jalisco, Mexico